CLINICAL TRIAL: NCT00094328
Title: An Open-label, Non-comparative, Multi-centre Study to Assess the Efficacy and Safety of Bicalutamide When Used in Combination With Anastrozole for the Treatment of Gonadotropin-independent Precocious Puberty in Boys With Testotoxicosis
Brief Title: Pediatrics Testotoxicosis Study [Bicalutamide Anastrozole Treatment for Testotoxicosis]
Acronym: BATT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6873C00047; BATT
Record Dates: First submitted 2004-10-16; First posted 2004-10-18 (Estimated); Results first posted 2009-07-09 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Puberty, Precocious
Keywords: Testotoxicosis; Familial Male-limited Precocious Puberty (FMPP)
MeSH Terms: conditions — Puberty, Precocious; Familial Testotoxicosis | interventions — bicalutamide; Anastrozole

ARMS (1):
- Bicalutamide with Anastrozole (Other): Bicalutamide in combination with Anastrozole
  Interventions: Drug: Bicalutamide; Drug: Anastrozole

INTERVENTIONS:
Drug: Bicalutamide — oral
  Other Names: Casodex
Drug: Anastrozole — oral
  Other Names: Arimidex; ZD1033

SUMMARY:
The primary objective of this study is to investigate whether bicalutamide given in combination with anastrozole once daily for 12 months is effective in treating testotoxicosis in boys. Testotoxicosis is a condition that causes early puberty in boys including growth in height, and development of muscles and sexual organs .

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent of parent/legal guardian and subject assent (as needed by local requirements)
* Male aged 2 years and over
* Diagnosis of testotoxicosis based on the following:
* Clinical features of Progressive sexual precocity documented by Tanner staging and evidence of symmetrical testicular enlargement
* Clinical features of significantly advanced bone age (defined as bone age of at least 12 months beyond chronological age)
* Pubertal levels of serum testosterone
* Prepubertal levels of serum gonadotropins
* Lack of an increase in serum gonadotropin levels following GnRH stimulation
* Other pathology excluded by:
* Undetectable plasma b human chorionic gonadotropin (bHCG). Samples with values below the LOQ will be reported as "<10 IU/L" which in the clinical setting equate to 'undetectable'.
* Normal levels of 17-hydroxyprogesterone (17-OHP)
* Normal levels of dehydroepiandrosterone sulphate (DHEAS)
* Naive to anti androgen receptor therapy:

(Note: Ketoconazole and Spironolactone are considered acceptable as is prior use of anastrozole or other aromatase inhibitors)

* A documented reliable height measurement taken > 6 months prior to study enrollment. Additionally for subjects who have previously received ketoconazole or spironolactone treatment, a documented reliable height measurement taken immediately prior to beginning this treatment.

(Note: for subjects who received such previous treatment only a single assessment is needed if it was taken immediately prior to beginning treatment and > 6 months prior to study entry)

* Subjects should be free of endocrine or other effects of previous treatment for testotoxicosis prior to study entry: to ensure this there should be 15 days or 4 drug half lives (whichever is the longer) washout period from prior medication for testotoxicosis.

Exclusion Criteria:

* Evidence of central precocious puberty as demonstrated by GnRH stimulation test
* Serum concentration of total or direct bilirubin, GGT, AST or ALT greater than 1.5 times the upper limit of normal for age
* Serum concentration of creatinine greater than 1.5 times the upper limit of normal for age
* Any concomitant medical condition that, in the opinion of the investigator, may expose a subject to an unacceptable level of safety risk or that affects subject compliance
* Known hypersensitivity to any of the study medications
* Participation in a clinical study at the time of enrollment

Ages: 2 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2004-11-22 (Actual); Primary Completion 2008-05-22 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri E Rukazenkov, MD, Study Director — AstraZeneca
Locations (15):
- United States (9):
  - Research Site, Birmingham, Alabama
  - Research Site, Jacksonville, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Minneapolis, Minnesota
  - Research Site, Tulsa, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Temple, Texas
  - Research Site, Spokane, Washington
- Research Site, London, Ontario, Canada
- Research Site, Montpellier, France
- India (2):
  - Research Site, Chennai
  - Research Site, New Dehli
- Research Site, Moscow, Russia
- Research Site, London, United Kingdom

REFERENCES:
- See also: CSR-D6873C00047.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=402&filename=CSR-D6873C00047.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 22 November 2004 and the last patient completed the 12 months visit on 7 May 2008. Patients were allocated treatment at 9 centres in 3 countries: India, the UK and the USA. Care for two patients, transferred from one US to a new approved US centre, therefore, patients were treated at 10 centres in total
Pre-assignment Details: Of the 24 patients enrolled, 10 failed eligibility criteria and were classed as screening failures while the remaining 14 patients were allocated treatment.
Groups:
- Open Label Bicalutamide With Anastrozole: Patients with testotoxicosis (familial male-limited precocious puberty) were given study drugs (bicalutamide in combination with anastrozole) orally once-daily for 12 months. The dosing of bicalutamide and anastrozole was independently tailored for each patient.
Period: Overall Study
Arm/Group | Open Label Bicalutamide With Anastrozole
Started | 14 (Received treatment)
Completed | 13 (Completed 12 months on treatment)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: Years] | 3.5 [2 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 12
  Race: Black | 1
  Race: Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic group: Hispanic/Latino | 1
  Ethnic group: African/American | 1
  Ethnic group: Asian | 3
  Ethnic group: Not Applicable | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Growth Rate (cm/Year)
Description: Change in growth rate after 12 months relative to the growth rate during the ≥6 month pre-study period, based on raw height data (cm/year).
Time Frame: Assessed after 12 months treatment
Population: All treated (AT) set
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 13
cm/year | -1.62 (5.13)
Statistical Analysis 1: Comparison: Open Label Bicalutamide With Anastrozole; The primary efficacy parameter, change in growth rate (cm/year) after 12 months relative to the baseline growth rate was analysed using a one sample t-test. A 95% 2-sided confidence interval was calculated for the mean change in growth rate; Test type: Other — One sample t-test; p = 0.278, t-test, 2 sided; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-4.72 to 1.48]

2. Primary Outcome: Change in Growth Rate (SD Units)
Description: Change in growth rate after 12 months relative to the growth rate during the ≥6 month pre-study period, calculated after adjustment for the chronological age of the patient (expressed as a standard deviation [SD] score).
Time Frame: Assessed after 12 months treatment
Population: All treated (AT) set
Measure: Mean (Standard Deviation); unit: SD units
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 13
SD units | -0.07 (1.78)
Statistical Analysis 1: Comparison: Open Label Bicalutamide With Anastrozole; The primary efficacy parameter, change in growth rate (SD units) after 12 months relative to the baseline growth rate was analysed using a one sample t-test. A 95% 2-sided confidence interval was calculated for the mean change in growth rate; Test type: Other — One sample t-test; p = 0.882, t-test, 2 sided; Median Difference (Final Values) = -0.07, 95% CI 2-sided [-1.15 to 1.00]

3. Secondary Outcome: Change in Growth Rate (cm/Year)
Description: Change in growth rate after 6 months of treatment relative to the growth rate during the ≥6 months pre-study period.
Time Frame: Assessed after 6 months treatment
Population: All treated (AT) set
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 13
cm/year | -0.70 (5.77)

4. Secondary Outcome: Change in Growth Rate (SD Units)
Description: Change in growth rate after 6 months of treatment relative to the growth rate during the ≥6 months pre-study period.
Time Frame: Assessed after 6 months treatment
Population: All treated (AT) set
Measure: Mean (Standard Deviation); unit: SD units
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 13
SD units | -0.14 (1.67)

5. Secondary Outcome: Change in Bone Age Maturation Rate (cm/Year)
Description: Radiographs were used to assess the bone age at ≥6 months pre-study, baseline, 6 and 12 months. The rate of change in bone age at baseline was calculated from a radiograph taken at least 6 months prior to study enrolment. The change in bone maturation after 6 months of treatment was calculated relative to the rate of change in bone age during the ≥ 6 months pre-study period.
Time Frame: Assessed after 6 and 12 months treatment
Population: Calculated on All treated analysis set for those patients who had a 6-month pre study radiograph.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 6
cm/year
  After 6 months treatment | -2.03 (0.38)
  After 12 months treatment | -2.29 (0.51)

6. Secondary Outcome: Change in Bone Age to Chronological Age Ratio
Description: Change in bone age to chronological age ratio after 6 and 12 months treatment relative to the baseline ratio for all patients.
Time Frame: Assessed after 6 and 12 months of treatment
Population: All treated (AT) set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 13
Ratio
  After 6 months treatment | -0.09 (0.14)
  After 12 months treatment | -0.24 (0.18)

7. Secondary Outcome: Number of Patients With Height Between 5th and 95th Percentile
Description: The number of patients whose height lies between the 5th and 95th percentiles (using the percentile tables on the WHO database) for chronological age at the 12 month assessment.
Time Frame: Assessed after 3, 6, 9 and 12 months of treatment
Population: All treated (AT) set
Measure: Number; unit: Participants
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 13
Participants
  After 3 months treatment | 3
  After 6 months treatment | 3
  After 9 months treatment | 3
  After 12 months treatment | 3

8. Secondary Outcome: Change in Predicted Adult Height (PAH)
Description: Radiographs are used to assess the bone age, the change in predicted adult height (PAH) is calculated from the bone age using the Bayley and Pinneau Method. The change in PAH is be calculated by subtracting the PAH at baseline from the PAH at 12 months.
Time Frame: Assessed after 12 months treatment
Population: Calculated on All treated analysis set, however, if bone age is less than 6 years or bone age is less than 7 years and bone age>=(chronological age-1) then PAH cannot be calculated using the Bayley and Pinneau method.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 9
cm | 6.21 (3.93)

9. Secondary Outcome: Change in Average Testicular Volume
Description: Testicular volume of both testes was measured using either ultrasound or an orchidometer. Testicular volume was measured at baseline and at 6 and 12 months. The change in testicular volume from baseline was calculated for the left and right testicle as well as the average across both testes by subtracting the baseline volume from the volumes at 6 and 12 months within each patient.
Time Frame: Assessed after 6 and 12 months of treatment
Population: All treated (AT) set
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Open Label Bicalutamide With Anastrozole
Number analyzed (Participants) | 13
mL
  After 6 months treatment | 1.46 (2.29)
  After 12 months treatment | 2.69 (2.51)

ADVERSE EVENTS:
Arm/Group | Open Label Bicalutamide With Anastrozole
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 13/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Bicalutamide With Anastrozole (N=14)
Abdominal Pain (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Asthenia (General disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Breast Tenderness (Reproductive system and breast disorders) | 2
Cafe Au Lait Spots (Skin and subcutaneous tissue disorders) | 1
Conjunctivitis (Eye disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Croup Infectious (Infections and infestations) | 2
Crying (Psychiatric disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Ear Infection (Infections and infestations) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gynaecomastia (Reproductive system and breast disorders) | 7
Headache (Nervous system disorders) | 3
Labyrinthitis (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Microcytosis (Blood and lymphatic system disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 2
Otitis Externa (Infections and infestations) | 1
Precocious Puberty (Endocrine disorders) | 6
Pyoderma (Infections and infestations) | 1
Pyrexia (General disorders) | 3
Respiratory Tract Infection Viral (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Seasonal Allergy (Immune system disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Staphylococcal Abscess (Infections and infestations) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Tonsillitis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Varicella (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to collaborate with AstraZeneca on the contents and formation of any publication or disclosure and to pay due consideration to comments and opinions offered. AstraZeneca have 60 days for final manuscript review and may require that submission for publication be delayed for a further 90 days in order to file patent applications.